CLINICAL TRIAL: NCT04952077
Title: MRI Biomarkers of Effective Tissue Reperfusion After Thrombectomy of an Acute Proximal Occlusion of the Anterior Circulation: MR-Reperfusion Longitudinal Study
Brief Title: MRI Biomarkers of Effective Tissue Reperfusion After Thrombectomy of an Acute Proximal Occlusion of the Anterior Circulation
Acronym: MR-Reperfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Liang LIAO, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A00716-35
Record Dates: First submitted 2021-06-17; First posted 2021-07-07 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Magnetic Resonance Imaging (MRI)

SUMMARY:
Cerebral infarction by proximal occlusion of the anterior circulation is common with major personal and societal consequences.

MRI is the gold standard for exploring stroke, especially ischemic, and a number of biomarkers on initial MRI (before reperfusion) are predictive of neurological prognosis. However, their spatiotemporal evolution in the suites of reperfusion is unclear.

Close monitoring by MRI would make it possible to precisely know the tissue, vascular and microvascular evolution of the infarct area and the penumbra after reperfusion, and thus to characterize MRI biomarkers associated with efficient tissue reperfusion.

The aim of the MR-Reperfusion study is to characterize new MRI biomarkers of efficient tissue reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 year-old
* Perfusion MRI assessment on admission;
* Admission for an acute infarction of the anterior circulation with proximal occlusion (tandem, distal internal carotid, or M1 segment of the middle cerebral artery);
* Initial mTICI = 0-1 on the initial angiography before treatment;
* Patient in complete autonomy (mRS ≤ 2) before the onset of symptoms;
* Mechanical thrombectomy (in combination or not with intravenous thrombolysis), within the first 6 hours of the onset of symptoms, or within 24 hours in case of clinical-radiological or radiological mismatch;
* Success of reperfusion estimated by an mTICI = 3 at the end of the procedure;
* Availability of MRI within 3 hours of angiographic reperfusion;
* To be able to understand the instructions given;
* Written consent given by the patient or a trusted person;
* To be enrolled in a social security plan;

Exclusion Criteria:

* Posterieur circulation obstruction;
* 3 months follow-up impossible with the completion of the MRI;
* Subject under a measure of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Description of MRI biomarkers (volume, location of the infarction and penumbra; collateral circulation; location, length of the thrombus; trans-cerebral, cortical venous changes) in patients with ischemic stroke successfully treated by thrombectomy | Admission to hospital, 3 hours, 24 hours, 7 days and 3 months after thrombectomy

SECONDARY OUTCOMES:
Kinetic evolution of MRI biomarkers (volume, location of the infarction and penumbra; collateral circulation; location, length of the thrombus; trans-cerebral, cortical venous changes) and its correlation with the functional prognosis (mRS score) | Admission to hospital, 3 hours, 24 hours, 7 days and 3 months after thrombectomy
Kinetic evolution of the NIHSS score and its correlation with the functional prognosis at 3 months evaluated by the mRS score. | Admission to hospital, 3 hours, 24 hours, 7 days and 3 months after thrombectomy
Description of MRI biomarkers (volume, location of the infarction and penumbra; collateral circulation; location, length of the thrombus; trans-cerebral, cortical venous changes) and its correlation with the hemorrhagic transformation (SWAN sequence) | 24 hours after thrombectomy
Radioclinical concordance evaluated by measuring MRI biomarkers (volume, location of the infarction and penumbra; collateral circulation; location, length of the thrombus; trans-cerebral, cortical venous changes), the mRS score and the NIHSS score | 3 months after thrombectomy

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France